CLINICAL TRIAL: NCT04638712
Title: Impact of (Neo)Adjuvant Therapy Associating Anthracyclines and Taxanes With or Without Trastuzumab on Skeletal Muscle in Breast Cancer Patients
Acronym: PROTECT-03
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Collaborators: UR 3072 - Mitochondries, Stress oxydant, Protection musculaire (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-006; 2020-A01266-33 (Other: IDRCB)
Record Dates: First submitted 2020-11-02; First posted 2020-11-20 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Body Composition; Quality of Life

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 without trastuzumab (Other)
  Interventions: Other: Microbiopsy sample; Other: Muscle echography, Maximal strength, Body composition, Quality of life and Physical activity level
- Group 2 with trastuzumab (Other)
  Interventions: Other: Microbiopsy sample; Other: Muscle echography, Maximal strength, Body composition, Quality of life and Physical activity level

INTERVENTIONS:
Other: Microbiopsy sample — before and after chemotherapy
Other: Muscle echography, Maximal strength, Body composition, Quality of life and Physical activity level — before and after chemotherapy

SUMMARY:
This is an interventional, prospective and monocentric study. This study includes the evaluation before and after (neo)adjuvant therapy of :

* one group of patients receiving anthracyclines and taxanes
* a second group of patients receiving anthracyclines, taxanes and trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

For group 1 without trastuzumab :

* Patients must be ≥ 18 years old
* Patients with breast cancer stage I to III
* Patients who will receive (neo)adjuvant anthracyclines and weekly taxane, without trastuzumab
* Patients must have a social security coverage
* Patients able to speak, read and understand French

For group 2 with trastuzumab :

* Patients must be ≥ 18 years old
* Patients with breast cancer grade I to III
* Patients who will receive (neo)adjuvant anthracyclines and weekly taxane, with trastuzumab
* Patients must have a social security coverage
* Patients able to speak, read and understand French

Exclusion Criteria:

* History of cancer
* Previous chemotherapy
* Patients with known chronic pathology (musculoskeletal disorders, autoimmune, vascular or neuromuscular disease)
* Pacemaker implantation
* Contraindication to physical condition evaluation
* Contraindication to local anesthesia required for microbiopsy
* Patients < 18 years old or patients ≥ 18 years old under guardianship, or supervision
* Psychiatric, musculoskeletal or neurologic disorders
* Women that are pregnant or breast-feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Change in vastus lateralis cross-sectional area | Between Week 18 and 24 after chemotherapy
  Measured from muscle microbiopsy sample

SECONDARY OUTCOMES:
Alteration of patients body composition | Baseline (=before chemotherapy) and Between Week 18 and 24 (=after chemotherapy)
  Assessment using bio-impedance analysis
Alteration of patients strength | Baseline (=before chemotherapy) and Between Week 18 and 24 (=after chemotherapy)
  Assessment of maximal isometric muscle strength for knee extensors measured with force sensors.
Alteration of patients muscle architecture | Baseline (=before chemotherapy) and Between Week 18 and 24 (=after chemotherapy)
  Assessment using muscle ultrasonography
Alteration of patients quality of life | Baseline (=before chemotherapy) and Between Week 18 and 24 (=after chemotherapy)
  Self-assessment questionnaire Functional Assessment of Cancer Therapy - General (FACT-G) (version 3)
Evaluation of patient cachexia | Baseline (=before chemotherapy) and Between Week 18 and 24 (=after chemotherapy)
  Questionnaire Functional Assessment of Anorexia/Cachexia Therapy (FAACT) (version 4)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Cancerologie Strasbourg Europe, Strasbourg, France

REFERENCES:
- [Result] Mallard J, Hucteau E, Hureau TJ, Pagano AF. Skeletal Muscle Deconditioning in Breast Cancer Patients Undergoing Chemotherapy: Current Knowledge and Insights From Other Cancers. Front Cell Dev Biol. 2021 Sep 14;9:719643. doi: 10.3389/fcell.2021.719643. eCollection 2021. PMID 34595171
- [Result] Mallard J, Hucteau E, Charles AL, Bender L, Baeza C, Pelissie M, Trensz P, Pflumio C, Kalish-Weindling M, Geny B, Schott R, Favret F, Pivot X, Hureau TJ, Pagano AF. Chemotherapy impairs skeletal muscle mitochondrial homeostasis in early breast cancer patients. J Cachexia Sarcopenia Muscle. 2022 Jun;13(3):1896-1907. doi: 10.1002/jcsm.12991. Epub 2022 Apr 4. PMID 35373507
- [Result] Mallard J, Hucteau E, Bender L, Charlot A, Debrut L, Pflumio C, Trensz P, Schott R, Favret F, Pivot X, Hureau TJ, Pagano AF. Development of skeletal muscle atrophy and intermuscular adipose tissue in patients with early breast cancer treated with chemotherapy. Am J Physiol Cell Physiol. 2022 Oct 1;323(4):C1325-C1332. doi: 10.1152/ajpcell.00373.2022. Epub 2022 Sep 12. PMID 36094434